CLINICAL TRIAL: NCT04613323
Title: Management of Thyroid Function in Hashimoto's Thyroiditis During Pregnancy: Real-word Experience in a Secondary Endocrine Centre in Italy
Brief Title: Management of Thyroid Function in Hashimoto's Thyroiditis During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centro Diagnostico Priamar (Other)
Responsible Party: Principal Investigator, Massimo Giusti, Associate Professor, Centro Diagnostico Priamar
Other Study IDs: Priamar001
Record Dates: First submitted 2020-07-14; First posted 2020-11-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2020-11

CONDITIONS: Hashimoto Disease; Pregnancy Related; Thyroid Dysfunction
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of thyroid function in pregnancy has been object of several guidelines in the last years. Normal thyroid function reduces prenatal and post-natal risks and gestational complaints. Trimester specific reference values of thyroid hormones and thyroid stimulating hormone (TSH) are available for selected geographic population but its are not yet are available in our country. Hashimoto's thyroiditis (HT) is the most frequent autoimmune thyroid disease which can induce thyroid dysfunction, mainly sub-clinical hypothyroidism. Due to the large incidence in women HT and its potential link with thyroid dysfunction this disease could be search and monitored before pregnancy. Anyway a strong recommendation is to test TSH levels in all patients seeking pregnancy at risk for thyroid dysfunction for a history or current symptoms/signs of thyroid dysfunction, known positivity od thyroid autoimmunity or goiter, a history of neck radiation, age >30 years, diabetes mellitus, previous infertility or pregnant loss, morbid obesity, living in area of moderate-severe iodine deficiency or recent administration of drugs/substance interfering with thyroid function.

DETAILED DESCRIPTION:
The aim of the study was to retrospectively evaluate from 2011 (data of publication of the first American Thyroid Association (ATA) guidelines for thyroid dysfunction in pregnancy) to now medical record of the a secondary level endocrine unit to verify the adherence to guidelines in the management of thyroid function in pregnant women with HT.

The investigators search

1. the adherence to clinical and biochemical endocrine evaluations before conception
2. the use (correct/un-correct) of L-T4 intervention and its monitoring
3. the difference in thyroid function control between women with a fix increment of- L-T4 posology (25 mcg/week more for each 2 kg increment in body weight) after the initial L-T4 adjustment or prescription
4. the clinical and biochemical endocrine evaluation 1-2 months after delivery
5. the outcome of pregnancy
6. the e-mail up-to-date survey on current of off-springs health

ELIGIBILITY:
Inclusion Criteria:

Adult HT pregnant women and adult pregnant women with nodular goiter with or whiteout previous known hypothyroidism.

Exclusion Criteria:

1. significant pre-pregnancy comorbidity including renal failure, severe liver disease, organ transplant, cardiac failure, psychiatric conditions requiring in-patient admission, history of eating disorder.
2. unable to have e-mail address
3. unavailable written consent
4. unable understand Italian language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult females in reproductive age
Study Population: Women with Hashimoto's thyroidis or/and gloiter
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Control of thyroid function in pregnancy | Through study completion, an average of 1 year
  Thyroid hormones and TSH

IPD SHARING:
Plan to Share IPD: No